CLINICAL TRIAL: NCT07268599
Title: Acoltremon Symptom Tracking and Relief Assessment in Moderate-to-Severe Dry Eye Disease
Brief Title: Moderate-to-Severe Dry Eye Disease Relief Using Acoltremon
Acronym: ASTRA
Status: Enrolling by invitation | Type: Observational
Sponsor: Colvard Kandavel Eye Center (Other)
Responsible Party: Principal Investigator, Ganesha Kandavel, Principal Investigator, Colvard Kandavel Eye Center
Other Study IDs: ASTRA-25859
Record Dates: First submitted 2025-11-21; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye Disease (DED)
Keywords: Dry Eye; Dry Eye Disease; Acoltremon
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Acoltremon — Patients will administer Acoltremon 0.003% as per labeled directions. Assessments with the Ocular Surface Disease Index (OSDI) will occur at Baseline, treatment at 14 days, and treatment at 28 days. Secondary endpoints include change from baseline rating scale 1-5 in severity of various symptoms of dry eye: Blurriness, eye irritation/Discomfort, Burning/Stinging, Photophobia/Pain, Sandy/gritty/Foreign Body Sensation, Fatigue/Tired Eyes).

SUMMARY:
To evaluate the impact of Acoltremon 0.003% on subjective dry eye symptoms using validated patient-reported outcome measures: Eye Dryness Score Visual Analog Scale (EDS-VAS). The primary aim is to characterize the rapidity of symptomatic relief in moderate to severe dry eye disease (DED), with attention to short-term therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older with clinical diagnosis of DED within past 6 months
* Use or desire for artificial tears for DED symptoms within past 2 months
* OSDI score >25 and <50 at Screening
* TBUT <10 seconds
* Baseline tCFS score ≥2 and ≤15 (modified NEI)

Exclusion Criteria:

* History of corneal or conjunctival surgery
* History of herpes zoster ophthalmicus, herpes simplex virus keratitis, or other viral corneal infection
* History of neurotrophic keratitis
* Prior significant facial trauma or sinus surgery
* Mental or physical condition impairing ability to complete questionnaires
* Use of Restasis®, Xiidra®, or Miebo within 30 days
* Use of other topical anti-inflammatory medications within 30 days
* Use of varenicline nasal spray within 30 days
* Use of artificial tears within 2 hours prior to screening or during study period
* Glaucoma requiring topical therapy
* Contact lens or eyelid scrub use within 7 days
* Punctal plugs within 14 days
* Oxervate historical use
* Amniotic membrane or Serum Tears historical use
* History of Sjögren's disease
* History of LASIK within 1 year

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Colvard-Kandavel Eye Center patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Ocular Surface Disease Index at 28 days | Baseline and 28 days
  Change from baseline in specific 1-5 categorical rating scale scoring at 28 days of dry eye symptoms: Blurriness, burning/stinging, eye irritation/discomfort, photophobia/pain, tired eyes/eye fatigue, sandy/gritty/foreign body sensation

CONTACTS AND LOCATIONS:
Overall Officials: Ganesha R Kandavel, MD, Principal Investigator — Colvard Kandavel Eye Center
Locations (1):
- Colvard-Kandavel Eye Center, Encino, California, United States

REFERENCES:
- [Background] Pucker AD, Ng SM, Nichols JJ. Over the counter (OTC) artificial tear drops for dry eye syndrome. Cochrane Database Syst Rev. 2016 Feb 23;2:CD009729. doi: 10.1002/14651858.CD009729.pub2. PMID 26905373
- [Background] Dry eye redefined: TFOS DEWS II report; 2017; 1-6. https://www.tfosdewsreport.org. Accessed 18 Feb 2022.
- [Background] Holland EJ, Luchs J, Karpecki PM, Nichols KK, Jackson MA, Sall K, Tauber J, Roy M, Raychaudhuri A, Shojaei A. Lifitegrast for the Treatment of Dry Eye Disease: Results of a Phase III, Randomized, Double-Masked, Placebo-Controlled Trial (OPUS-3). Ophthalmology. 2017 Jan;124(1):53-60. doi: 10.1016/j.ophtha.2016.09.025. Epub 2016 Oct 27. PMID 28079022
- [Background] Bacharach J, Kannarr SR, Verachtert A, Gupta PK, Razeen M, Cavet ME, Vittitow JL, Lang J, Chester TM, Ziemanski JF, White DE. Early Effects of Perfluorohexyloctane Ophthalmic Solution on Patient-Reported Outcomes in Dry Eye Disease: A Prospective, Open-Label, Multicenter Study. Ophthalmol Ther. 2025 Apr;14(4):693-704. doi: 10.1007/s40123-025-01097-z. Epub 2025 Feb 22. PMID 39985746
- [Background] Wirta DL, Galor A, Aune CA, Vollmer PM, Liang E, Meides AS, Krosser S. Long-Term Safety and Efficacy of a Water-Free Cyclosporine 0.1% Ophthalmic Solution for Treatment of Dry Eye Disease: ESSENCE-2 OLE. Cornea. 2024 May 21;44(6):692-700. doi: 10.1097/ICO.0000000000003567. PMID 38771801
- [Background] Wolffsohn JS, Arita R, Chalmers R, Djalilian A, Dogru M, Dumbleton K, Gupta PK, Karpecki P, Lazreg S, Pult H, Sullivan BD, Tomlinson A, Tong L, Villani E, Yoon KC, Jones L, Craig JP. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017 Jul;15(3):539-574. doi: 10.1016/j.jtos.2017.05.001. Epub 2017 Jul 20. PMID 28736342
- [Background] Miller KL, Walt JG, Mink DR, Satram-Hoang S, Wilson SE, Perry HD, Asbell PA, Pflugfelder SC. Minimal clinically important difference for the ocular surface disease index. Arch Ophthalmol. 2010 Jan;128(1):94-101. doi: 10.1001/archophthalmol.2009.356. PMID 20065224
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Stonecipher KG, Torkildsen GL, Ousler GW 3rd, Morris S, Villanueva L, Hollander DA. The IMPACT study: a prospective evaluation of the effects of cyclosporine ophthalmic emulsion 0.05% on ocular surface staining and visual performance in patients with dry eye. Clin Ophthalmol. 2016 May 13;10:887-95. doi: 10.2147/OPTH.S101627. eCollection 2016. PMID 27257373
- [Background] Uchino M, Schaumberg DA. Dry Eye Disease: Impact on Quality of Life and Vision. Curr Ophthalmol Rep. 2013 Jun;1(2):51-57. doi: 10.1007/s40135-013-0009-1. PMID 23710423
- [Background] Friedman NJ. Impact of dry eye disease and treatment on quality of life. Curr Opin Ophthalmol. 2010 Jul;21(4):310-6. doi: 10.1097/ICU.0b013e32833a8c15. PMID 20467319
- [Background] Craig JP, Nelson JD, Azar DT, Belmonte C, Bron AJ, Chauhan SK, de Paiva CS, Gomes JAP, Hammitt KM, Jones L, Nichols JJ, Nichols KK, Novack GD, Stapleton FJ, Willcox MDP, Wolffsohn JS, Sullivan DA. TFOS DEWS II Report Executive Summary. Ocul Surf. 2017 Oct;15(4):802-812. doi: 10.1016/j.jtos.2017.08.003. Epub 2017 Aug 8. PMID 28797892